CLINICAL TRIAL: NCT01303055
Title: Multicenter Trial on Effects of Alogliptin on Pancreatic Beta Cell Function
Brief Title: Effects of Alogliptin on Pancreatic Beta Cell Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aichi Gakuin University (Other)
Responsible Party: Takahiro Tosaki, Aichi Gakuin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGU-248
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pancreatic beta Cell; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Metformin; Hypoglycemic Agents; Physiological Effects of Drugs; Pharmacologic Actions; hemoglobin A1c protein, human; Oral Glucose Tolerance Test
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — alogliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alogliptin (Experimental): Alogliptin 25 mg
  Interventions: Drug: Alogliptin
- Metformin (Active Comparator): Metformin 750 mg
  Interventions: Drug: Metformin 750 mg

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily : two years
  Other Names: Nothing
  Arms: Alogliptin
Drug: Metformin 750 mg — Metformin 750 mg, tablets, orally, thrice daily: two years
  The dose increase is possible up to its maximum, 2250 mg, so that HbA1c is maintained below 6.9 %.
  Other Names: Nothing
  Arms: Metformin

SUMMARY:
It is reported that pancreatic beta cell function is already declined at pre-diabetic stage, impaired glucose tolerance (IGT). It has not been clarified whether inhibitors of the dipeptidyl peptidase IV enzyme (DPP-IV inhibitors) improve beta cell function on human pancreas, however, if efficacy is ensured, they may become the first medicine to be chosen for treatments of type 2 diabetes and IGT.

In this trial, a DPP-IV inhibitor, Alogliptin, or Metformin are given to diabetic patients whose HbA1c level is below 7.9%. Oral glucose tolerance test (OGTT) will be conducted before, a year after, and two years after the beginning of the trial and beta cell function will be evaluated.

DETAILED DESCRIPTION:
Patients will be randomly allocated to two groups. They will receive either Alogliptin or Metformin.

Alogliptin: The investigators will start with 25 mg QD and the dose will be maintained.

Metformin: The investigators will start with 250 mg QD and the dose will be slowly increased to 750 mg TID. The dose increase is possible up to its maximum, 2250 mg, so that HbA1c is maintained below 6.9%. However, increase in dose with elder patients requires careful consideration.

Participants taking part in this study will receive dietary and exercise coaching. Participation in this study is expected to last up to 2 years.

Patients will terminate from the trial when their HbA1c exceeds 8.4% for more than three months.

The investigators will evaluate beta cell function by conducting 75 g OGTT before, a year after, and two years after the beginning of the trial. Alogliptin or Metformin will be stopped three days before the OGTT. The investigators will make sure that urine ketone is negative before an oral glucose load.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as type 2 diabetes with HbA1c level below 7.9% and haven't received oral hypoglycemic agents or insulin treatments for the past three months.

Exclusion Criteria:

* Patients whose 75 g OGTT 30-minutes insulin secretion exceeds 100 μU/ml
* Patients with renal failure with serum creatinine level ≧ 1.2
* Patients with hepatocirrhosis
* Patients with proliferative diabetic retinopathy or worse
* Patients with acute infectious disease
* Patients who are treated with steroids
* Patients with cancer
* Pregnant patients
* Patients with malfunction of the heart (NYHA classification III-IV)
* Patients who are decided to be inappropriate subjects by study physicians

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
beta cell function evaluated from 75 g OGTT | 2 years
  75 g OGTT: glucose level, blood insulin level, c-peptide immunoreactivity (pre-test, 30 mins, 60 mins, 120 mins), fasting blood proinsulin
  Oral glucose tolerance test ( OGTT ) will be conducted before, a year after, and two years after the beginning of the trial.

SECONDARY OUTCOMES:
1,5-AG level | 2 years
  Secondary end points include HbA1c level.

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Tosaki, MD, PhD, Study Chair — Aichi Gakuin University
Locations (4):
- Japan (4):
  - Dept. of Intern. Med., School of Dentistry, Aichi Gakuin University, Nagoya, Aichi-ken
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya, Aichi-ken
  - Diabetes Clinic, Okazaki East Hospital, Okazaki, Aichi-ken
  - Diabetes Center, Yokkaichi Social Insurance Hospital, Yokkaichi, Mie-ken